CLINICAL TRIAL: NCT03028051
Title: Chronic Pain, Life Style Factors and Quality of Life
Status: Completed | Type: Observational
Sponsor: Helsinki University Central Hospital (Other)
Responsible Party: Principal Investigator, Tarja Heiskanen, MD, Ph.D., pain specialist, Helsinki University Central Hospital
Other Study IDs: KROKIETA
Record Dates: First submitted 2017-01-02; First posted 2017-01-23 (Estimated); Last update posted 2017-01-25 (Estimated); Status verified 2017-01

CONDITIONS: Chronic Pain
MeSH Terms: conditions — Chronic Pain

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Blood samples frozen for possible further biochemical analysis (vitamin D, S-PTH, S-TSH, cytokines, P-Ca++)
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- chronic pain patients: Finnish speaking, adult chronic pain patients, aged 18 - 75 years, referred to pain clinic

SUMMARY:
Chronic pain, life style factors and quality of life (KROKIETA) is a multicenter study that aims to analyze life style factors, socioeconomic and psychometric properties, metabolic problems, drug use, quality of life and biochemical variables in chronic non-cancer pain patients. The life style factors will be compared to those of normal population. At baseline, the study patients fill in questionnaires (A-E), the patients´ weight, length, waist and blood pressure are measured, pain-related factors are recorded and blood samples taken. Changes in the quality of life of the study patients will be evaluated by questionnaires during follow-up at 2 years and 5 years.

DETAILED DESCRIPTION:
Chronic pain co-occurs with risk factors for cardiovascular diseases, depression, smoking and sleep problems. Nutrition and low physical activity may predispose to chronic pain. To gain information on the life style factors of adult chronic pain patients referred to university hospital or central hospital pain clinics in Finland, 477 patients have been recruited to the study. The patients fill in questionnaires on sociodemographic factors, pain, medication, use of health services, physical activity, smoking, use of alcohol or other substances, sleep, quality of life, nutrition and psychological factors at their first visit to the pain clinic. Height, weight, waist circumference, blood pressure and pulse are measured by the study nurse. A blood sample for analysis of blood sugar, cholesterol (total, LDL, HDL), triglycerides, HbA1c and sensitive C-reactive protein (CRP) is taken. The pain clinician records the pain diagnosis, medication and other methods of pain management chosen. The patients will be sent follow-up questionnaires at 2 years and 5 years after baseline.

ELIGIBILITY:
Inclusion Criteria:

* age 18 to 75 years
* chronic non-cancer pain
* Finnish-speaking
* referred to a multidisciplinary pain management center

Exclusion Criteria:

* inability to fill in questionnaires in Finnish
* cancer pain

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult, Finnish-speaking patients, aged 18-75 years, referred to a pain clinic for multidisciplinary pain treatment.
Sampling Method: Non-Probability Sample
Enrollment: 477 (Actual)
Dates: Start 2014-09; Primary Completion 2016-12 (Actual); Study Completion 2016-12 (Actual)

PRIMARY OUTCOMES:
Change of quality of life as assessed by 15 Dimensions questionnaire between baseline and 2 years | 2 years
  Baseline and 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Eija Kalso, Professor, Principal Investigator — Helsinki University Central Hospital

IPD SHARING:
Plan to Share IPD: No